CLINICAL TRIAL: NCT02640430
Title: A Preliminary Randomized Trial of the FreeAspire Versus PEP-bottle After Acute Exacerbation in COPD Patients With Mucus Hypersecretion and Decreased Cough Efficiency.
Brief Title: Randomized Trial of the FreeAspire Versus PEP-bottle After Acute Exacerbation in COPD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maugeri Foundation (Other)
Responsible Party: Principal Investigator, Andrea Zanini, MD, Maugeri Foundation
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: maugerifoundation
Record Dates: First submitted 2015-12-17; First posted 2015-12-29 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- standard treatment (Active Comparator): Control group will be made of 20 COPD patients with severe and very severe airflow obstruction, mucus hypersecretion and reduced cough efficiency referred to standard pulmonary rehabilitation after acute exacerbation.
  Control group will b treated with PEP-bottle over 10 daily sessions (20 minutes twice a day). Patients are asked to breath against a positive expiratory pressure determined by a column of water in a bottle (PEP Bolltle). PEP is one of the validated treatment used in the clearance of bronchial secretions in COPD patients.
  All patients will receive regular treatment with inhaled bronchodilators and inhaled steroids according to current guidelines for their disease stage. Each patient will sign an informed consent form.
  Interventions: Device: standard treatment
- Free Aspire (Experimental): Experimental group will be made of 20 COPD patients with severe and very severe airflow obstruction , mucus hypersecretion , and reduced cough efficiency referred to standard pulmonary rehabilitation after acute exacerbation.
  Patients are asked to use FREE ASPIRE Free Aspire is an electro-medical device which removes bronchopulmonary secretions noninvasively, without using a suction catheter and without generating airway pressure, positive or negative.
  All patients will receive regular treatment with inhaled bronchodilators and inhaled steroids according to current guidelines for their disease stage. Each patient will sign an informed consent form.
  Interventions: Device: Free Aspire

INTERVENTIONS:
Device: standard treatment — 20 minutes, twice a day for 10 sessions
  Other Names: PEP bottle
  Arms: standard treatment
Device: Free Aspire — 20 minutes, twice a day for 10 sessions
  Arms: Free Aspire

SUMMARY:
BACKGROUND: Studies have shown that COPD patients with bronchial hypersecretion have increased risk of acute exacerbations. FREE ASPIRE is an electro-medical device which removes bronchopulmonary secretions noninvasively, without using a suction catheter and without generating airway pressure.

AIM: To compare FREE ASPIRE activity with the traditional treatment using PEP-bottle in the clearance of bronchial secretions in COPD patients METHODS: Forty severe and very severe COPD patients with mucus and reduced cough will be evaluated. Group comparison will be made between Intervention group using VAKÜM system (Free Aspire®), and Control group using traditional treatment with PEP-bottle over 10 daily sessions (20 minutes twice a day). Primary outcomes are changes in arterial blood gases exchanges, in perceived dyspnea and in symptom of bronchial encumbrance.

EXPECTED RESULTS: A higher significant reduction of the perceived dyspnea and of perceived bronchial encumbrance is supposed in the Intervention group. Additional benefits among the secondary outcomes are also hypothesized in the same group.

DETAILED DESCRIPTION:
Background. Chronic obstructive pulmonary disease (COPD) is a complex and heterogeneous disease, whose pathophysiological aspects remain still today unknown. Among the various phenotypes, chronic bronchitis presents mucus hypersecretion as clinical distinctive character, having also a pathogenic role. Studies have shown that COPD patients with bronchial hypersecretion have increased risk of acute exacerbations. This risk has a negative impact on disease progression, quality of life of patients and direct and indirect costs. It is necessary to identify more efficient instruments and techniques that allow to obtain airway clearance, usable in most clinical settings, including rehabilitation centers, and suitable for the largest number of patients. FREE ASPIRE is an electro-medical device which removes bronchopulmonary secretions noninvasively, without using a suction catheter and without generating airway pressure, positive or negative. FREE ASPIRE uses a VAKÜM technology , by accelerating expiratory flow of airways, and it can also be used in patients with reduced cough efficiency.

Aim of the study. To compare FREE ASPIRE activity with the traditional treatment using PEP-bottle in the clearance of bronchial secretions in COPD patients with mucus hypersecretion and decreased cough efficiency, and to test the hypothesis that the newly developed VAKÜM technology may provide additional clinical benefits over conventional treatment in terms of clinical and functional outcomes.

Materials and methods. This is a single center, randomized and preliminary prospective study. The study has been approved by the Internal Review Board of the Malcantonese Hospital, 6980 Castelrotto, Switzerland and the procedures will be performed in the Division of Internal and Respiratory Medicine. Following a preliminary run-in period, group comparison will be made between Intervention group using VAKÜM system (Free Aspire, MPR, Legnano, Italy), and Control group using traditional treatment with PEP-bottle over 10 daily sessions (20 minutes twice a day). All patients will receive regular treatment with inhaled bronchodilators and inhaled steroids according to current guidelines for their disease stage. Each patient will sign an informed consent form. Considering a probability of 15% drop-out rate of randomized patients, we consider to enroll at least 24 patients per group.

Spirometric lung volumes, respiratory muscle strength (MIP and MEP), arterial blood gases, perceived dyspnea (by BDI-TDI scale), peak expiratory air flows (PEF and PCEF), perceived bronchial encumbrance (by VAS scale) and quality of life (Clinical COPD Questionnaire, CCQ, CAT) will be recorded in both groups pre-to-post PR.

Continuous data will be reported as mean ± standard deviation (SD), unless otherwise specified. The distribution of variables will be assessed by means of Kolmogorov-Smirnov Goodness-of-Fit test. Comparisons between quantitative and qualitative variables will be determined by paired and unpaired t test, and χ2 test, when appropriate. Relationships between variables will be assessed by the Pearson's correlation coefficient (r) and the Spearman's correlation coefficient (rs), when appropriate. Data analyses and graphical presentations will be performed using GraphPad Prism 5 (GraphPad Software, San Diego, California, USA) and SPSS version 20 (IBM, Armonk, New York, USA). A p-value < 0.05 will be considered as statistically significant.

Study start date: January 2016 Estimated study completion date: June 2017 Expected results. A higher significant reduction of the perceived dyspnea and of perceived bronchial encumbrance is supposed in the Intervention group. Additional benefits among the secondary outcomes are also hypothesized in the same group.

ELIGIBILITY:
Inclusion Criteria:

COPD patients with:

* severe and very severe airflow obstruction (FEV1<50%)
* mucus hypersecretion (sputum production >30 ml/die)
* reduced cough efficiency (Peak Cough Expiratory Flow > 160 and < 300 l/min)

Exclusion Criteria:

* Any medical or psychological condition that in opinion of the investigator influences the ability to follow the programme

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10; Primary Completion 2018-10 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
perceived symptom of bronchial encumbrance | 10 days
  VAS Scale

SECONDARY OUTCOMES:
changes in arterial blood gases exchanges | 10 days
  BGA
perceived dyspnea | 10 days
  BDI-TDI
changes in peak expiratory air flows | 10 days
  PFT
lung volumes | 10 days
  PFT
respiratory muscle strength | 10 days
  MIP-MEP

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Spanevello, MD, Study Director — Maugeri Foundation
Locations (2):
- Maugeri Foundation, Tradate, VA, Italy
- Division of Internal and Respiratory Medicine, Ospedale Malcantonese, Fondazione Giuseppe Rossi, Castelrotto, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
publication

REFERENCES:
- [Background] Bellone A, Lascioli R, Raschi S, Guzzi L, Adone R. Chest physical therapy in patients with acute exacerbation of chronic bronchitis: effectiveness of three methods. Arch Phys Med Rehabil. 2000 May;81(5):558-60. doi: 10.1016/s0003-9993(00)90034-0. PMID 10807091
- [Background] Osadnik CR, McDonald CF, Jones AP, Holland AE. Airway clearance techniques for chronic obstructive pulmonary disease. Cochrane Database Syst Rev. 2012 Mar 14;2012(3):CD008328. doi: 10.1002/14651858.CD008328.pub2. PMID 22419331
- [Background] Vestbo J, Hurd SS, Agusti AG, Jones PW, Vogelmeier C, Anzueto A, Barnes PJ, Fabbri LM, Martinez FJ, Nishimura M, Stockley RA, Sin DD, Rodriguez-Roisin R. Global strategy for the diagnosis, management, and prevention of chronic obstructive pulmonary disease: GOLD executive summary. Am J Respir Crit Care Med. 2013 Feb 15;187(4):347-65. doi: 10.1164/rccm.201204-0596PP. Epub 2012 Aug 9. PMID 22878278
- [Background] Prescott E, Lange P, Vestbo J. Chronic mucus hypersecretion in COPD and death from pulmonary infection. Eur Respir J. 1995 Aug;8(8):1333-8. doi: 10.1183/09031936.95.08081333. PMID 7489800